CLINICAL TRIAL: NCT01650597
Title: A Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-42165279 in Healthy Male Subjects
Brief Title: A Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-42165279 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR100707; 42165279EDI1001 (Other: Janssen-Cilag International NV); 2011-002861-39 (EudraCT Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2014-05

CONDITIONS: Healthy Volunteers; Pharmacokinetics
Keywords: Healthy volunteers; Pharmacokinetics; Free fatty amides
MeSH Terms: interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 - Panel 1 (Experimental): The participants will receive 3 or 4 ascending doses (2.5, 10, 30, 100, 250, 500 mg) of JNJ-42165279 and placebo during the study.
  Interventions: Drug: JNJ-42165279 2.5 - 500 mg oral; Drug: Placebo
- Part 1 - Panel 2 (Experimental): The participants will receive 3 or 4 ascending doses (2.5, 10, 30, 100, 250, 500 mg) of JNJ-42165279 and placebo during the study.
  Interventions: Drug: JNJ-42165279 2.5 - 500 mg oral; Drug: Placebo
- Part 2 (parallel)- additional cohort (Experimental): The participants will receive repeated daily dosing of 100 mg JNJ-42165279 or placebo for 6 consecutive days.
  Interventions: Drug: Placebo; Drug: JNJ-42165279 100 mg oral

INTERVENTIONS:
Drug: JNJ-42165279 2.5 - 500 mg oral — Type=exact number, unit=mg, numbers=2.5, 10, 30, 100, 250 and 500, form=suspension, route=oral use. One single dose administered orally.
  Arms: Part 1 - Panel 1; Part 1 - Panel 2
Drug: Placebo — Type=exact number, unit=mg, form=solution, route=oral use. One single dose administered orally.
Drug: JNJ-42165279 100 mg oral — Type=exact number, unit=mg, form=solution, route=oral use. One single dose administered orally.
  Arms: Part 2 (parallel)- additional cohort

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of single ascending doses as well as repeated doses of JNJ-42165279 in healthy male participants.

DETAILED DESCRIPTION:
This is a single-site, randomized (participants are assigned to treatment by chance), double-blind study (neither physician nor participant knows whether the participant is receiving active treatment or placebo). Placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect. This study consists of two parts (part 1, single dosing and part 2, multiple dosing). Part 1: An alternating panel design will be used, whereby the first panel of 9 participants will receive the first, third, and fifth administered doses, while the second panel of 9 participants will receive the second, fourth, and sixth administered doses.Up to 2 additional dosings (1 per panel) may be evaluated to further understand the study drug. For each dose administration, 6 participants will be assigned to active treatment and 3 to placebo. Each participant will receive JNJ-42165279 on 2 occasions and placebo once during the first 3 dosings. The planned doses of JNJ-42165279 range from 2.5 to 500 mg. The sponsor and investigator will review blinded data associated with each dose prior to administration of the next dose. Participants will check into the study center the morning prior to each dosing (Day -1) and will remain at the center until discharge 72 hours after dosing (Day 4). Participants will be dosed approximately every 4 weeks. Part 2: A separate cohort of 9 healthy male volunteers will receive repeated daily dosing of 100 mg JNJ-42165279 or placebo (6 participants will receive JNJ-42165279 and 3 participants will receive placebo) for 6 consecutive days. Participants will check into the study center the morning prior to their first dosing (Day -1) and will remain at the center until discharge 72 hours after receiving their last dose on Day 6. Participants in Part 1 and 2 will return for a follow-up visit 7 to 14 days after their final discharge from the study center.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index between 18 and 30 kg/m2 and body weight not less than 50 kg.
* Must adhere to required contraception (subject and partner, if applicable) during the study and for 3 months after study
* Must agree to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Has history of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, recent surgery or trauma.
* Has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Has clinically significant abnormal values for hematology, clinical chemistry, coagulation, or urinalysis at screening or at first admission to the study center.
* Has clinically significant abnormal physical examination, neurological examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or at first admission to the study center. Subjects with a QTcF interval >450 msec or QRS interval ≥110 msec will be excluded.
* Has use of any prescription or nonprescription medications or herbal supplements, except for paracetamol, within 14 days before the first dose of study drug. Paracetamol is not allowed within 1 day (Day -1) before the first dose of study drug.
* Has known allergy, hypersensitivity, or intolerance to hypromellose (the excipient of JNJ-42165279)
* Has Known allergy to heparin or history of heparin induced thrombocytopenia
* Has positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B core antibody (HBcAB), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV)
* Has history of significant drug or alcohol abuse within past 5 years, or has a positive drug screen
* Smoking or use of nicotine-containing substances within past 2 months
* Blood donation or blood loss within past 3 months
* Recent use of an investigational drug or device

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidents of adverse events amongst participants (Part 1) | Day -21 to Day 114 (~19 wks)
  As a measure of safety.
Incidents of adverse events amongst participants (Part 2) | Day -21 to Day 23 (~6 wks)
Pharmacokinetics of JNJ-42165279 as measured by Cmax (Part 1) | Day 1 to Day 4
  Cmax is defined as maximum plasma concentration of JNJ-42165279.
Pharmacokinetics of JNJ-42165279 as measured by Cmax (Part 2) | Day 1 to Day 7
Pharmacokinetics of JNJ-42165279 as measured by AUC (Part 1) | Day 1 to Day 4
  AUC is defined area under the plasma concentration time curve from 0 to t hours post dosing of JNJ-42165279.
Pharmacokinetics of JNJ-42165279 as measured by AUC (Part 2) | Day 1 to Day 7

SECONDARY OUTCOMES:
Fatty acid amide hydrolase (FAAH) inhibition in white blood cells (WBCs) (Part 1) | Day 1 to Day 4
FAAH inhibition in WBC (Part 2) | Day 1 to Day 7 and Day 9
Effects on mood (Part 1) | Day 1 and Day 2
  This is measured by scores on Patient Reported Outcome (PRO) questionnaires (Profile of Mood States [POMS], State version of the State-Trait Anxiety Inventory [STAIS], and the Exercise-Induced Feeling Inventory [EFI]). The POMS is a valid and reliable self-report scale that can be utilized to assess both positive and negative, transient, fluctuating mood states. The STAIS is a commonly-used, validated instrument to assess anxiety. The EFI assesses emotions commonly associated with exercise.
Effects on mood (Part 2) | Day 1 to Day 9
Effects on cognition (Part 1) | Day -1 and Day 1
  This is assessed by the time to complete Trail Making Test (TMT).
Effects on cognition (Part 2) | Day -1, Day 1 and Day 6
Effects on pain tolerance (Part 1) | Day -1 to Day 2
  This is measured by pressure pain tolerance threshold using an electronic pressure algometer.
Effects on drowsiness (Part 2) | Day 1 to Day 6
  This is measured by Stanford Sleepiness Scale (SSS). This 7 point Likerttype scale is used to rate the drowsiness with the descriptors ranging from "feeling active, vital, alert, and wide awake" (score= 1) to "no longer fighting sleep, sleep onset soon, and having dream like thoughts" (score=7).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Principal Investigator — Janssen-Cilag International NV
Locations (1):
- Merksem, Belgium